CLINICAL TRIAL: NCT04721574
Title: The Effect of Bright Light Therapy on Sleep and Quality of Life in Patients
Brief Title: Bright Light Therapy on Post-stroke Insomniawith Post-stroke Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Wonhyoung Kim, Professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-05-005
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Stroke Sequelae
MeSH Terms: interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright light therapy (Active Comparator): Daily exposure to a high brightness LED light box for 30 minutes as soon as possible after awakening, preferably between 7 and 8 AM in the patient's hospital room The device emits 10,000 lux of cool-white fluorescent light at 50-75 cm from the screen to the cornea with an ultraviolet filter
  Interventions: Device: Philips EnergyUp Energy light HF3418/01
- Sham Therapy (Sham Comparator): Light-therapy with filters that reduced lamp output to less than 50 lux. for 30 minutes as soon as possible after awakening.
  Interventions: Device: Philips EnergyUp Energy light HF3418/01 with filter

INTERVENTIONS:
Device: Philips EnergyUp Energy light HF3418/01 — high brightness LED light box
  Other Names: Bright light therapy
  Arms: Bright light therapy
Device: Philips EnergyUp Energy light HF3418/01 with filter — high brightness LED light box with filters that reduced lamp output to less than 50 lux
  Other Names: Bright light therapy with filter
  Arms: Sham Therapy

SUMMARY:
The objective of this study was to determine the effectiveness of bright light therapy as a treatment for early, mild-to-moderate stroke patients with post-stroke insomnia.

ELIGIBILITY:
Inclusion Criteria:

* first occurrence of stroke for the patient
* matched International Classification of Diseases (ICD)-10 codes (nontraumatic subarachnoid hemorrhage [I60], nontraumatic intracerebral hemorrhage [I61], other and unspecified nontraumatic intracranial hemorrhage [I62], or cerebral infarction [I63]) (World Health Organization, 1997)
* mild-to-moderate stroke (the National Institutes of Health Stroke Scale ≤14)
* age ≥18 years
* satisfactory cognitive function
* post-stroke insomnia.

Exclusion Criteria:

* Mini Mental State Examination (MMSE) score of ≤10
* recurrent stroke
* aphasia
* transient ischemic attack
* schizophrenia, bipolar disorder, mood disorder, previous insomnia disorder, or dementia before stroke
* taking sleeping pills or antidepressants for 5 or more days within a 6-month timespan before the onset of stroke
* post-stroke delirium
* a National Institutes of Health Stroke Scale score ≥ 14
* previous eye disease or post-stroke eye disease
* severe auditory impairment
* the use of psychotropic medications (hypnotics, benzodiazepine, benzodiazepine agonists, antidepressants [mirtazapine or trazodone] or antipsychotics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
total sleep duration in actigraphy | 4 weeks
  the sum [in minutes] of all sleep epochs between sleep onset and sleep end
sleep onset latency in actigraphy | 4 weeks
  the interval between time-to-bed and sleep onset
sleep efficiency in actigraphy | 4 weeks
  (SE%, the percentage of time spent asleep while in bed
wake after sleep onset in actigraphy | 4 weeks
  sum [in minutes] of all awake epochs between sleep onset and sleep end
number of awakenings in actigraphy | 4 weeks
  number of awakenings

SECONDARY OUTCOMES:
the insomnia severity index | 4 weeks
  Subjective sleep parameters, 0-28, higher scores indicate more acute symptoms of insomnia
the Pittsburgh Sleep Quality Index | 4 weeks
  Subjective sleep parameters, 0-21, higher scores indicate more poor sleep quality
The Epworth Sleepiness Scale | 4 weeks
  Subjective sleep parameters, 0-24, 0-28, higher scores indicate more daytime sleepiness
the Fatigue Severity Scale | 4 weeks
  Subjective sleep parameters, 0-36, 0-28, higher scores indicate greater fatigue.
The Patient Health Questionnaire-9 | 4 weeks
  depression, 0-27, higher scores indicate more severe of depression.
The generalized Anxiety Disorder-7 | 4 weeks
  anxiety, 0-21, higher scores indicate more severe of anxiety
The World Health Organization Quality of Life Scale Abbreviated Version | 4 weeks
  overall quality of life through self-reporting, with four subscales in overall health: physical health, psychological health, social relationships, and environmental health. The higher sum in each subscale signified better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Inha university hospital, Incheon, Jung-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim WH, Joa KL, Kim CB, Lee HS, Kang SG, Jung HY, Bae JN. The Effect of Bright Light Therapy on Sleep and Quality of Life in Patients With Poststroke Insomnia. Psychosom Med. 2022 Jan 1;84(1):123-130. doi: 10.1097/PSY.0000000000001014. PMID 34581703